CLINICAL TRIAL: NCT04923724
Title: Impact on Tourniquet Use on Functional Outcomes and Complications After TKA
Brief Title: Tourniquet on Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201805014
Record Dates: First submitted 2021-05-19; First posted 2021-06-11 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Arthritis Knee
MeSH Terms: interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: Patients are put into 2 study groups. One group gets a tourniquet during surgery and one group does not.
Who Masked: Participant
Masking Description: Participants do not know which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tourniquet during surgery (Active Comparator): Patients in this group get a tourniquet during surgery.
  Interventions: Device: tourniquet
- No Tourniquet during surgery (Active Comparator): Patients in this group do not get a tourniquet during surgery.
  Interventions: Device: No tourniquet

INTERVENTIONS:
Device: tourniquet — tourniquet is a device used during total knee surgery.
  Arms: Tourniquet during surgery
Device: No tourniquet — tourniquet is a device used during total knee surgery, this group does not get one
  Arms: No Tourniquet during surgery

SUMMARY:
The purpose of this study is determine the effect on novel pressure-regulating tourniquet use on pain, functional recovery, sleep and total blood loss following total knee arthroplasty.

DETAILED DESCRIPTION:
Functional recovery after total knee arthroplasty (TKA) has seen dramatic improvement over the past 20 years through advances in surgical technique, implant design, perioperative pain management strategies, and physical therapy protocols. Tourniquet use during TKA, however, remains controversial due to conflicting reports in the literature on these benefits and risks of its use. Reported advantages of tourniquet use include improved visualization of the surgical field and decreased intraoperative blood loss. Reported disadvantages of tourniquet use include increased postoperative pain and slower functional recovery as a direct result of the pressure of the tourniquet on the thigh during the procedure.

Traditionally with tourniquet use during TKA, the limb is exsanguinated and the tourniquet is raised to a fixed, pressure at the beginning of the case, typically 250mmHg to 350mmHg, and let down after closure. A novel tourniquet design that adjusts the tourniquet pressure in real-time based on intraoperative patient blood pressure measurements. This design may allow for the tourniquet to be inflated at a lower mean pressure while still maintaining efficacy.

A prospective study comparing total blood loss, pain and functional recovery after TKA using this novel tourniquet design, design (Zimmer A.T.S.® 4000TS Automatic Tourniquet System, with disposable contour cuffs) and TKA without tourniquet would further the current literature. Total blood loss will be calculated by previously validated methods. Pain and functional recovery will be closely monitored throughout the postoperative period using a patient wearable activity tracker (FitBit Inspire HR) and a smartphone-based patient engagement platform with integrated digital surveys paired with smart-brace based home PT assessments (FocusMotion).Pain and functional recovery will be closely monitored throughout the postoperative period using a patient wearable activity tracker (FitBit Inspire HR) and a smartphone-based patient engagement platform with integrated digital surveys paired with smart-brace based home PT assessments (FocusMotion). Applying this technology to the proposed study can help identify problematic pain that is not appreciable during admission; given the fact that markers of inflammation and myocyte damage increase over time until at least post-operative day 3, it is possible that TKAs performed under tourniquet may have pain and narcotic requirements not appreciated with short-stay admissions . The proposed study will further the literature on pain and narcotic use in the early time period after TKA, and will help identify if tourniquet has an effect on these variables.

Furthermore, sleep quality is a component of functional recovery and is correlated with pain. Knee osteoarthritis affects general quality of life by increasing sleep disturbance and nighttime wakening, and this is correlated with the pre-operative radiographic severity of disease. Sleep quality is affected in the immediate post-operative period after TKA as well, but improves by 3-6 months post-operatively . The proposed study would be the largest prospective study investigating the effect of TKA on pain and sleep quality, as well as being the first to investigate tourniquet use as a factor affecting sleep quality and pain. The proposed study would be the first to collect both subjective and objective data on the subject, using validated survey measurements as well as the data collected by the Fitbit Inspire HR device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and up
* Primary unilateral TKA
* BMI<45
* Primary diagnosis of osteoarthritis
* Patient has a iOS or Android smartphone capable of running FitBit and FocusMotion applications

Exclusion Criteria:

* Revision TKA
* Bilateral TKA
* Pregnancy
* Prisoners
* Pre-existing functionally-limiting neurologic disorder
* Narcotic dependence, defined as oxycodone/hydrocodone use >5days/week
* History of unprovoked VTE/PE
* Inability to complete baseline functional testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Barrack, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Creve Coeur, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery
Started | 82 | 83
Completed | 57 | 58
Not Completed | 25 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 39 | 82
  >=65 years | 14 | 19 | 33
Age, Continuous [Mean (Full Range); unit: years] | 63.4 [18 to 80] | 64.6 [18 to 80] | 64 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 34 | 56
  Male | 35 | 24 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 57 | 58 | 115

OUTCOME MEASURES:

1. Primary Outcome: Pain After TKA Measured by VAS Pain Survey on Focusmotion App
Description: Effect of tourniquet use on pain after TKA, 0-10 scale with 10 being higher pain, VAS pain survey
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery
Number analyzed (Participants) | 58 | 57
score on a scale | 2.8 (1.5) | 2.6 (1.8)

2. Secondary Outcome: Functional Recovery Measured by Oxford Knee Score Scale
Description: Effect of tourniquet use on functional recovery after TKA. Score each question (item) from 0 to 4 with 0 being the worst outcome and 4 being the best outcome. The scores are then summed to produce an overall score running from 0 (worst possible) to 48 (best outcome).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery
Number analyzed (Participants) | 58 | 57
score on a scale | 43.0 (6.28) | 41.37 (8.84)

3. Secondary Outcome: Functional Recovery Measured by Forgotten Joint Score
Description: Effect of tourniquet use on functional recovery after TKA. Scale measures how much patient is aware of their joint after surgery.
  a total of 12 questions are answered asking about awareness of the knee joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. Final score = 100 - ((sum(item01 to item12) - 12)/48*100) 0:Represents the worst possible score, indicating the highest level of joint awareness and the least ability to forget.
  100:Represents the best possible score, indicating the lowest level of joint awareness and the greatest ability to forget
Time Frame: 1 year
Population: not all patients completed this survey, that is why the numbers are inconsistent with other surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery
Number analyzed (Participants) | 47 | 40
score on a scale | 68.4 (28.2) | 70.9 (77.4)

4. Secondary Outcome: Functional Recovery Measured by Normal Knee Survey
Description: Effect of tourniquet use on functional recovery after TKA measured by a score of 0-100, 100 being knee feels normal, 0 means knee does not feel normal
Time Frame: 1 year
Population: not all patients completed this survey, that is why participant numbers are inconsistent with other surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery
Number analyzed (Participants) | 45 | 39
score on a scale | 79.3 (90) | 81.5 (20.1)

5. Other Pre Specified Outcome: Hours of Sleep Per Night Postoperatively
Description: Investigate sleep quality in post-operative period after TKA using fitbit tracker average hours of sleep at night
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: hours of sleep
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery
Number analyzed (Participants) | 41 | 28
hours of sleep | 5.41 (2.23) | 6.47 (1.63)

6. Other Pre Specified Outcome: Total Blood Loss
Description: effect of tourniquet use on total calculated blood loss after TKA. this is calculated by change in hemoglobin in g/dL from preop to periop.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: g/dL hemoglobin
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery
Number analyzed (Participants) | 54 | 53
g/dL hemoglobin | 13.9 (1.4) | 11.5 (1.3)

ADVERSE EVENTS:
Time Frame: Ae's collected up to 1 year.
Description: the adverse events were not caused by the study
Arm/Group | Tourniquet During Surgery | No Tourniquet During Surgery
All-Cause Mortality (participants affected / at risk) | 1/57 | 0/58
Serious Adverse Events (participants affected / at risk) | 1/57 | 0/58
Other Adverse Events (participants affected / at risk) | 0/57 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tourniquet During Surgery (N=57) | No Tourniquet During Surgery (N=58)
urinary retention lower abdominal and back pain (Hepatobiliary disorders) | 1 (1) | 0 (0) — patient had urinary retention and had to stay in hospital

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT04923724/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT04923724/ICF_001.pdf